CLINICAL TRIAL: NCT02154854
Title: Effect of Advagraf on Arterial Stiffness and on Vascular Fibrosis Plasma Markers on de Novo Renal Transplant Patients
Brief Title: Prospective Study to Measure Vascular Parameters (Ancillary Study of ADEQUATE)
Acronym: ADEQUATEartère
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Tours (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PHAO2011/YL/ADEQUATE-A; 2011-003184-29 (EudraCT Number)
Record Dates: First submitted 2014-05-27; First posted 2014-06-03 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-05

CONDITIONS: De Novo Transplant Disease
Keywords: Renal; Transplantation; Tacrolimus; Arterial stiffness; Vascular fibrose plasma markers

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A - tacrolimus half-dose (Experimental): Immunosuppressive strategy with 50 % reduction of Advagraf® daily dose at M4 (randomization) and unchanged MMF dose. Targeted tacrolimus trough level are to be higher than 3 ng/mL . If the dose is not in adequation with the dispensable units, the prescribed dose will be the closest higher dose.
  Drug: Tacrolimus targeted half-dose
  Interventions: Drug: Tacrolimus targeted half-dose
- Group B - tacrolimus unchanged dose (Experimental): Immunosuppressive strategy will remain identical after randomization (M4): unchanged Advagraf® and MMF doses. Targeted tacrolimus trough level are to be between 7 and 12 ng/mL Drug: Tacrolimus targeted plain dose
  Interventions: Drug: Tacrolimus targeted plain dose

INTERVENTIONS:
Drug: Tacrolimus targeted half-dose
  Other Names: Advagraf®
  Arms: Group A - tacrolimus half-dose
Drug: Tacrolimus targeted plain dose
  Other Names: Advagraf®
  Arms: Group B - tacrolimus unchanged dose

SUMMARY:
The purpose of this study is to compare parallel-group effects between 4 months and 12 months post-transplantation 2 values of target residual concentrations of Advagraf on vascular parameters in de novo renal transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 et 70 years
* Patient accepting to give a written informed consent
* Recipients of a first renal allograft (deceased or living, non HLA identical donor with compatible ABO blood type)
* Randomized in the ADEQUATE study
* Patients must have at J112 +/- 3 days a stable renal function (MDRD 4) with an absence of DSA since transplantation.
* Negative T cross-match in cytotoxicity
* Tolerate a daily dose of MMF at 1g

Exclusion Criteria:

* Acute rejection during the first months
* Existence of a BK infection since M3
* Proteinuria/reatininuria ratio > 1g/g since M3

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2013-07; Primary Completion 2015-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Aorta stiffness at one year post-tranplantation | 12 months
  Evaluate the aorta stiffness at 1 year post-renal transplantation and its evolution in patients who received a half reduction of their daily dose of Advagraf ® 4 months after transplantation compared with patients whose dose has not been divided.

SECONDARY OUTCOMES:
Blood pressure | 12 months
  Evaluate peripheral and central blood pressures, the impact of reflected pressure waves and coupling cardiocirculatory (on the functional plan) and evaluate endothelial activation, factors promoting the vascular fibrosis and oxidant stress level (on biological plan) at 1 year post-renal transplantation and their evolution in patients who received a hal reduction of their daily dose Advagraf ® to four months of the transplant when compared with patients whose dose was not divided.
Endothelial activation at one year post-tranplantation | 12 months
  Evaluate peripheral and central blood pressures, the impact of reflected pressure waves and coupling cardiocirculatory (on the functional plan) and evaluate endothelial activation, factors promoting the vascular fibrosis and oxidant stress level (on biological plan) at 1 year post-renal transplantation and their evolution in patients who received a hal reduction of their daily dose Advagraf ® to four months of the transplant when compared with patients whose dose was not divided.

CONTACTS AND LOCATIONS:
Overall Officials: Robinson JOANNIDES, Principal Investigator — University Hospital, Rouen
Locations (11):
- France (11):
  - CHU de Amiens, Amiens
  - CHU de Angers, Angers
  - CHU de Caen, Caen
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - HEGP, Paris
  - Necker, Paris
  - CHU de Rennes, Rennes
  - CHU de Rouen, Rouen
  - CHU de Strasbourg, Strasbourg
  - CHU de Toulouse, Toulouse
  - CHRU de Tours, Tours